CLINICAL TRIAL: NCT02343640
Title: Ultrasound Study of Season-Long Joint Changes to College Baseball Players
Status: Completed | Type: Observational
Sponsor: California State University, Northridge (Other)
Responsible Party: Principal Investigator, Johnathan Anthony Erb, Student, California State University, Northridge
Other Study IDs: 1415-093
Record Dates: First submitted 2015-01-14; First posted 2015-01-22 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Complete Tear Ulnar Collateral Ligament
Keywords: Baseball; Ulnar collateral ligament

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Baseball players: Members of the baseball team, both pitchers and fielders, who participate in repetitive baseball throwing and are exposed to damage of the ulnar collateral ligament in the arm that is used for throwing.

SUMMARY:
The purpose of this study is to use ultrasound imaging to determine if there are certain frequencies, durations, and intensities of baseball pitching that expose a college baseball player to increased risk of injury to their ulnar collateral ligament of their elbow throughout one baseball season.

DETAILED DESCRIPTION:
This study aims to use ultrasound imaging to assess the health of the ulnar collateral ligament (UCL) of the elbow, which acts as a major stabilizer in overhead throwing athletes and is often injured in baseball pitchers. The health of the UCL will be assessed by measured the amount of laxity in the UCL, identified as the distance between the end of the humerus (arm bone) where the UCL originates and the beginning of the ulna (forearm bone) where the UCL ends. An increase in this distance indicates an increase in laxity of the ligament, which is a risk factor for injury/tearing of the ligament with repetitive throwing seen in baseball pitchers. Measurements will be made at rest and under 3 pounds of valgus stress at 30 degrees of elbow flexion where the UCL acts as the main stabilizer of the elbow. Valgus stress is necessary for this procedure because damage to the ligament will be most clearly seen in this position when compared to the measurement at rest.

Measurements will be made to both the right and left elbows, as well as both the right and left knees. The purpose of including the knees in this protocol is so that the subjects are blinded to the true intention of the study. Due to the psychological harm that could occur if the subjects know the focus of the study is their UCL, the study will be presented to the subjects such that the research team is viewing all structures within the elbow and knee, and their overall flexibility, strength, and bony changes will be monitored throughout the season using ultrasound. Therefore, the ultrasound measurements of the knee will be sham measurements, and only measurements made at the elbow will be recorded.

In addition to ultrasound, measurements of range of motion will be performed at each testing session. Motions to be tested will be: shoulder flexion, extension, abduction, internal rotation, and external rotation; elbow flexion and extension; wrist flexion and extension; hip flexion, extension, abduction, internal rotation, and external rotation; knee flexion and extension. Recent studies have found significant results for deficits in range of motion correlating to UCL tears, so this data will be used in conjunction with measurements of laxity of the UCL as seen with ultrasound.

Ultrasound imaging and range of motion testing will be performed on the same 10 subjects four times throughout one baseball season: before the first game of the season, after 20 games have been played, after 40 games have been played, and after the last game of the season has been played. During this period, pitching data will be collected and recorded for each pitcher. Data to be collected includes number of pitches thrown, number of each type of pitch thrown, number of innings pitched, velocity of all pitches, time in days between pitching appearances.

ELIGIBILITY:
Inclusion Criteria:

* Must be a member of the CSU Northridge baseball team
* Able to provide written, informed consent
* Understand instruction in English
* Be between the age of 18 and 24 years

Exclusion Criteria:

* Is not a member of the CSU Northridge baseball team
* Experience pain or injury during testing procedures of the research study

Ages: 18 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Members of the CSU Northridge baseball team
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Joint distance | 18 weeks
  Allows for a measurement of distance, in millimeters, of the UCL from the humerus to the ulna to be made using ultrasound imaging.

SECONDARY OUTCOMES:
Goniometry | 18 weeks
  Measures the available amount of motion, in degrees, at multiple joints.

CONTACTS AND LOCATIONS:
Overall Officials: Johnathan A Erb, Principal Investigator — CSU Northridge; Aimie Kachingwe, Study Director — CSU Northridge

REFERENCES:
- [Background] Ciccotti MG, Atanda A Jr, Nazarian LN, Dodson CC, Holmes L, Cohen SB. Stress sonography of the ulnar collateral ligament of the elbow in professional baseball pitchers: a 10-year study. Am J Sports Med. 2014 Mar;42(3):544-51. doi: 10.1177/0363546513516592. Epub 2014 Jan 28. PMID 24473498
- [Background] Ciccotti MC, Hammoud S, Dodson CC, Cohen SB, Nazarian LN, Ciccotti MG. Stress ultrasound evaluation of medial elbow instability in a cadaveric model. Am J Sports Med. 2014 Oct;42(10):2463-9. doi: 10.1177/0363546514542805. Epub 2014 Aug 14. PMID 25125692
- [Background] Sasaki J, Takahara M, Ogino T, Kashiwa H, Ishigaki D, Kanauchi Y. Ultrasonographic assessment of the ulnar collateral ligament and medial elbow laxity in college baseball players. J Bone Joint Surg Am. 2002 Apr;84(4):525-31. doi: 10.2106/00004623-200204000-00003. PMID 11940610
- [Background] Smith W, Hackel JG, Goitz HT, Bouffard JA, Nelson AM. Utilization of sonography and a stress device in the assessment of partial tears of the ulnar collateral ligament in throwers. Int J Sports Phys Ther. 2011 Mar;6(1):45-50. PMID 21655456
- [Background] Nazarian LN, McShane JM, Ciccotti MG, O'Kane PL, Harwood MI. Dynamic US of the anterior band of the ulnar collateral ligament of the elbow in asymptomatic major league baseball pitchers. Radiology. 2003 Apr;227(1):149-54. doi: 10.1148/radiol.2271020288. Epub 2003 Feb 28. PMID 12616000
- [Background] Harada M, Takahara M, Sasaki J, Mura N, Ito T, Ogino T. Using sonography for the early detection of elbow injuries among young baseball players. AJR Am J Roentgenol. 2006 Dec;187(6):1436-41. doi: 10.2214/AJR.05.1086. PMID 17114533
- [Background] Wilk KE, Macrina LC, Fleisig GS, Aune KT, Porterfield RA, Harker P, Evans TJ, Andrews JR. Deficits in glenohumeral passive range of motion increase risk of elbow injury in professional baseball pitchers: a prospective study. Am J Sports Med. 2014 Sep;42(9):2075-81. doi: 10.1177/0363546514538391. Epub 2014 Jun 18. PMID 24944295
- [Background] Davidson PA, Pink M, Perry J, Jobe FW. Functional anatomy of the flexor pronator muscle group in relation to the medial collateral ligament of the elbow. Am J Sports Med. 1995 Mar-Apr;23(2):245-50. doi: 10.1177/036354659502300220. PMID 7778713
- [Background] Anz AW, Bushnell BD, Griffin LP, Noonan TJ, Torry MR, Hawkins RJ. Correlation of torque and elbow injury in professional baseball pitchers. Am J Sports Med. 2010 Jul;38(7):1368-74. doi: 10.1177/0363546510363402. Epub 2010 Apr 16. PMID 20400752
- [Background] Wilk KE, Macrina LC, Fleisig GS, Porterfield R, Simpson CD 2nd, Harker P, Paparesta N, Andrews JR. Correlation of glenohumeral internal rotation deficit and total rotational motion to shoulder injuries in professional baseball pitchers. Am J Sports Med. 2011 Feb;39(2):329-35. doi: 10.1177/0363546510384223. Epub 2010 Dec 4. PMID 21131681
- [Background] Dines JS, Frank JB, Akerman M, Yocum LA. Glenohumeral internal rotation deficits in baseball players with ulnar collateral ligament insufficiency. Am J Sports Med. 2009 Mar;37(3):566-70. doi: 10.1177/0363546508326712. Epub 2008 Dec 4. PMID 19059890
- [Background] Garrison JC, Cole MA, Conway JE, Macko MJ, Thigpen C, Shanley E. Shoulder range of motion deficits in baseball players with an ulnar collateral ligament tear. Am J Sports Med. 2012 Nov;40(11):2597-603. doi: 10.1177/0363546512459175. Epub 2012 Sep 26. PMID 23019251
- [Background] Bushnell BD, Anz AW, Noonan TJ, Torry MR, Hawkins RJ. Association of maximum pitch velocity and elbow injury in professional baseball pitchers. Am J Sports Med. 2010 Apr;38(4):728-32. doi: 10.1177/0363546509350067. Epub 2010 Jan 21. PMID 20093420
- [Background] Aguinaldo AL, Chambers H. Correlation of throwing mechanics with elbow valgus load in adult baseball pitchers. Am J Sports Med. 2009 Oct;37(10):2043-8. doi: 10.1177/0363546509336721. Epub 2009 Jul 24. PMID 19633230
- [Background] Posner M, Cameron KL, Wolf JM, Belmont PJ Jr, Owens BD. Epidemiology of Major League Baseball injuries. Am J Sports Med. 2011 Aug;39(8):1676-80. doi: 10.1177/0363546511411700. Epub 2011 Jun 27. PMID 21709023
- [Background] Conte S, Requa RK, Garrick JG. Disability days in major league baseball. Am J Sports Med. 2001 Jul-Aug;29(4):431-6. doi: 10.1177/03635465010290040801. PMID 11476381
- [Background] Azar FM, Andrews JR, Wilk KE, Groh D. Operative treatment of ulnar collateral ligament injuries of the elbow in athletes. Am J Sports Med. 2000 Jan-Feb;28(1):16-23. doi: 10.1177/03635465000280011401. PMID 10653538
- [Background] Podesta L, Crow SA, Volkmer D, Bert T, Yocum LA. Treatment of partial ulnar collateral ligament tears in the elbow with platelet-rich plasma. Am J Sports Med. 2013 Jul;41(7):1689-94. doi: 10.1177/0363546513487979. Epub 2013 May 10. PMID 23666850